CLINICAL TRIAL: NCT05413772
Title: Practical Use of Temocillin in Enterobacteriaceae Resistant to Third Generation of Cephalosporins: Experience of Two French University Hospitals
Brief Title: Temocillin in ESBL-Enterobacteriaceae Infections
Acronym: TMO2016
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210920
Record Dates: First submitted 2022-01-24; First posted 2022-06-10 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-11

CONDITIONS: Infectious Disease
Keywords: extended-spectrum-β-lactamase-producing Enterobacteriaceae; carbapenem-sparing agent; urinary tract infection; bacteraemia; temocillin
MeSH Terms: conditions — Communicable Diseases; Urinary Tract Infections; Toxemia | interventions — temocillin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Temocillin received empirically: Temocillin received in probabilistic , in curative context or in preventive use (prophylaxis)
  Interventions: Other: Temocillin
- Temocillin received on second line of treatment: Temocillin received second-line therapy in curative context or in preventive use (prophylaxis)
  Interventions: Other: Temocillin

INTERVENTIONS:
Other: Temocillin — To evaluate the clinical course of patients who received temocillin. To evaluate the efficacy and safety of temocillin in different situations Enterobacteriaceae ESBL infections

SUMMARY:
Because of the increasing incidence of infections with multi-drug resistant enterobacteriaceae, we need alternative treatments to spare carbapenems. Temocillin could be an interesting option but its position is only defined for the curative treatment of urinary tract infections. We would like to explore others indications comparing two groups : one using temocillin empirically for treatment or prophylaxis and the second using it in second line whatever the indication is.

DETAILED DESCRIPTION:
We will retrospectively include every patient who received at least 24 hours of temocillin for the treatment of an extended-spectrum beta-lactamase Enterobacteriaceae (ESBL-E) infection from January to December 2016 in two university hospitals (centres 1 and 2). Each treatment indication will be recorded including off-label prescriptions. Patients will be classified in 2 treatment groups: group 1 received a probabilistic antibiotherapy first (3GC or carbapenem or piperacillin/tazobactam or fluoroquinolones) followed by temocillin as second line treatment. Group 2 was defined by the use of temocillin as first line treatment or as prophylaxis.

Data collection : Clinical, biological and pharmaceutical data will be retrieved from medical chart. The patient's referring physician and/or the department will be contacted for further information on missing data. Remote outcomes will be retrieved either by hospital records if the patient is rehospitalized in the meantime or by contacting directly the patient by phone or e-mail. Demographic characteristics, comorbidities, type and location of infection, treatment, side effects, biological results, follow-up duration, treatment and outcome will be collected. For all antibiotics, doses, route and scheme administration, duration, first, second and third line of antibiotic (after temocillin) will be retrieved from medical chart.

Case definition and outcome: Treatment failure in curative use is defined by the persistence of clinical symptoms 72h after starting the antibiotic and/or clinical worsening leading to a switch to broad-spectrum antibiotic and/or recurrence of initial symptoms and/or identification of the same bacterial species with the same susceptibility pattern as initially observed (same or new location). Treatment failure in prophylactic use is defined by the persistence of the enterobacteria according to the indication of prophylaxis (e.g. urine). All deaths and lost-to-follow-up will be considered as failures (worst case scenario). Treatment success is defined by the absence of failure in the four weeks after treatment. We will use the Sequential Organ Failure Assessment (SOFA) score in predicting mortality in patients with ESBL-E infections included in our study.

Microbiological definitions : The susceptibility of the isolates to temocillin wil be determined by disc diffusion method (Biorad®, Marnes-la-Coquette, France) according to the guidelines of the CA-SFM ("Comité de l'Antibiogramme - Société Française de Microbiologie", Antibiogram Committee - French Society of Microbiology ). The Minimum Inhibitory Concentration (MIC) of temocillin will be determined by E-test (bioMérieux®, Marcy l'Étoile, France) on Mueller-Hinton agar using the manufacturer's instructions. MIC results will be also interpreted according to the 2016 guidelines of the CA-SFM.18

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* All patients who received at least 24 hours of temocillin for the treatment of ESBL enterobacteriaceae infection / colonization from January to December 2016 in the university hospitals of Tenon and Pitié Salpêtrière. All indications, including excluding recommendations.
* Informed and not opposed to the use of their data

Exclusion Criteria:

* Patient < 18 years
* Pregnancy
* Refusal to participate
* Multi-resistant bacterial infection not treated with temocillin
* Temocillin resistant bacteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18, hospitalized in any department from 01/01/16 to 12/15/16 at CHU Pitié-Salpêtrière or CHU Tenon, having received at least 24 hours of temocillin for an ESBL enterobacteria infection / colonization whatever or the indication.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Number of patients with failure or success | 10 days
  Definition of failure: persistence of clinical symptoms 72h after starting the antibiotic and/or clinical worsening (ie : fever, cough, sputum, urinary symptoms, diarrhea...) leading to a switch to broad-spectrum antibiotic and/or recurrence of initial symptoms and/or identification of the same bacterial species, retrieved in collection samples, with the same susceptibility pattern as initially observed (same or new location)

SECONDARY OUTCOMES:
Number of patients with treatment related adverse events as assessed by CTCAE v6.0 | 28 days
  Any side effect described in the medical file : Clostridium difficile colitis, renal failure, rash, for example.
  Collection of information in the medical file in order to explore the reason of failure : analyse of others potential failure's causes (other cause of fever for example)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Bonnet, MD, Principal Investigator — Pitie-Salpetriere University Hospital; Sophie Vimont, MD, Principal Investigator — Tenon Hospital
Locations (2):
- France (2):
  - Pitié-Salpêtrière University Hospital, Paris
  - Tenon University Hospital, Paris

IPD SHARING:
Plan to Share IPD: No